CLINICAL TRIAL: NCT01708720
Title: Safety and Immunogenicity of Sabin-IPV and Adjuvanted Sabin-IPV in Healthy Adults
Brief Title: Safety and Immunogenicity of a New Inactivated Polio Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pauline Verdijk (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor-Investigator, Pauline Verdijk, Clinical Research Scientist, National Institute for Public Health and the Environment (RIVM)
Organization: National Institute for Public Health and the Environment (RIVM) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NVI-256A; 2010-024581-22 (EudraCT Number)
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Poliomyelitis
Keywords: Vaccination; Inactivated Poliomyelitis Vaccine; Polio; Sabin
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sabin-IPV (Experimental): Single intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 20, 32, and 64 D-antigen units respectively of Sabin-1,-2 and -3 per dose
  Interventions: Drug: Sabin-IPV
- Adjuvanted Sabin-IPV (Experimental): Single intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 10, 16, and 32 D-antigen units respectively of Sabin-1,-2 and -3 per dose, adjuvanted with 0.5 mg aluminium hydroxide
  Interventions: Drug: Adjuvanted Sabin-IPV
- IPV (Active Comparator): Single intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 40, 8, and 32 D-antigen units respectively of Mahoney, MEF-1 and Saukett poliovirus per dose
  Interventions: Drug: IPV

INTERVENTIONS:
Drug: IPV
  Other Names: Inactivated poliomyelitis vaccine; Inactivated polio vaccine; Inactivated poliovirus vaccine
  Arms: IPV
Drug: Sabin-IPV
  Arms: Sabin-IPV
Drug: Adjuvanted Sabin-IPV
  Arms: Adjuvanted Sabin-IPV

SUMMARY:
The purpose of this trial is to determine whether the new inactivated polio vaccine that is based on attenuated poliovirus strains is safe and to evaluate the immune response in healthy adults.

DETAILED DESCRIPTION:
The goal of this study is to assess the safety and immunogenicity of Sabin-IPV and adjuvanted Sabin-IPV produced with the production process set up for technology transfer by the National Institute for Public Health and the Environment (RIVM, formerly the Netherlands Vaccine Institute (NVI).

* The primary objective is to evaluate safety (local and systemic reactions) of intramuscular injection with Sabin-IPV and adjuvanted Sabin-IPV in healthy adults (first in human).
* The secondary objective is to evaluate immunogenicity of Sabin-IPV and adjuvanted Sabin-IPV in healthy immunized adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 49, inclusive at the time of enrolment
* in good health as determined by the outcome of medical history, physical examination screening/baseline labs and clinical judgment of the investigator
* Male
* Must have received polio vaccinations with OPV according to the Polish National Immunization Program as a child based on vaccination cards or information given by subjects during interview with investigator
* Preferred: number (and date) of polio vaccinations known
* Willingness and ability to adhere to the study regimen
* Having a signed informed consent form

Exclusion Criteria:

* IPV or OPV booster dose after the age of 12 years
* Positive for HIV, Hepatitis B or Hepatitis C
* Known or suspected allergy against any of the vaccine components
* History of unusual or severe reactions to any previous vaccination
* Known or suspected disease or use of medication that may influence the immune system
* Known or suspected immune deficiency
* Systemic treatment with corticosteroids within one month before screening
* Administration of plasma (including immunoglobulins) or blood products three months prior to the study
* Blood donation within one month before screening
* Any vaccination within three months before screening and during the study until the last visit
* History of any neurological disorder including epilepsy or febrile seizures
* Evidence of excessive alcohol use or drug use
* Any infectious disease at the time of screening and/or inclusion
* Participation in another clinical trial within three months before screening
* Abnormal pre-treatment laboratory parameters which are clinically relevant according to the investigator
* Bleeding disorders or the usage of anticoagulants

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse reactions following vaccination | 4 days or until adverse reactions have resolved

SECONDARY OUTCOMES:
Level of virus neutralizing titers in serum | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Verdijk, PhD, Study Director — Institute for Public Health and the Environment
Locations (1):
- Szpital Internistyczny cetrum Badan Farmakologii Klinicznej Monipol Sp. z o.o., Krakow, Poland

REFERENCES:
- [Background] Bakker WA, Thomassen YE, van't Oever AG, Westdijk J, van Oijen MG, Sundermann LC, van't Veld P, Sleeman E, van Nimwegen FW, Hamidi A, Kersten GF, van den Heuvel N, Hendriks JT, van der Pol LA. Inactivated polio vaccine development for technology transfer using attenuated Sabin poliovirus strains to shift from Salk-IPV to Sabin-IPV. Vaccine. 2011 Sep 22;29(41):7188-96. doi: 10.1016/j.vaccine.2011.05.079. Epub 2011 Jun 7. PMID 21651934
- [Background] Verdijk P, Rots NY, Bakker WA. Clinical development of a novel inactivated poliomyelitis vaccine based on attenuated Sabin poliovirus strains. Expert Rev Vaccines. 2011 May;10(5):635-44. doi: 10.1586/erv.11.51. PMID 21604984
- [Result] Verdijk P, Rots NY, van Oijen MG, Oberste MS, Boog CJ, Okayasu H, Sutter RW, Bakker WA. Safety and immunogenicity of inactivated poliovirus vaccine based on Sabin strains with and without aluminum hydroxide: a phase I trial in healthy adults. Vaccine. 2013 Nov 12;31(47):5531-6. doi: 10.1016/j.vaccine.2013.09.021. Epub 2013 Sep 21. PMID 24063976